CLINICAL TRIAL: NCT00027443
Title: Giant Cell Myocarditis Treatment Trial Pilot Study
Brief Title: Study of Muromonab-CD3 and Cyclosporine in Patients With Giant Cell Myocarditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-1986-01; FD-R-001986-0
Record Dates: First submitted 2001-12-05; First posted 2001-12-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-10

CONDITIONS: Myocarditis
Keywords: Giant Cell Myocarditis
MeSH Terms: conditions — Myocarditis | interventions — Muromonab-CD3; Cyclosporine

INTERVENTIONS:
Drug: Muromonab-CD3
Drug: Cyclosporine

SUMMARY:
This is a study to determine the efficacy of muromonab-CD3 and cyclosporine as treatment in patients with giant cell myocarditis (GCM). T lymphocytes appear to be involved in GCM. Muromonab-CD3 has been shown to reduce the number of lymphocytes and cyclosporine inhibits lymphocyte activation. This treatment may prolong patient survival until transplantation or ventricular assist device placement is possible.

DETAILED DESCRIPTION:
Each patient will be randomized to receive either standard care and immunosuppression therapy (treatment group) or standard care alone (control group). To prevent bias, randomization will be stratified by recency of symptom onset to ensure that both the treatment and control groups are balanced with respect to it. Within each of these 2 strata, permuted-block randomization will be done to keep the number of treatment and control patients balanced. Due to the necessary monitoring of the patients randomized to receive immunosuppression therapy, treatment cannot be blinded. Approximately 1 year after the last patient has been randomized, the observed times from randomization to the composite endpoint (death, transplantation, or LVD placement) will be compared in the treatment and control groups.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Idiopathic heart failure and/or arrhythmia of less than 3 months duration
* Endomyocardial biopsy diagnostic of idiopathic giant cell myocarditis
* Negative pregnancy test

Exclusion criteria:

* Clinical evidence of sepsis or active infection (e.g., meningitis or osteomyelitis)
* Pregnant
* Any contraindication to immunosuppression
* Allergy to cyclosporine or muromonab-CD3
* Creatinine greater than 2.5 mg/dL
* AST or ALT greater than 3 times upper limit of normal
* Other severe concurrent disease that would preclude study
* Unreliable or uncooperative subject

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-08; Study Completion 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Leslie T Cooper, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cooper LT Jr, Hare JM, Tazelaar HD, Edwards WD, Starling RC, Deng MC, Menon S, Mullen GM, Jaski B, Bailey KR, Cunningham MW, Dec GW; Giant Cell Myocarditis Treatment Trial Investigators. Usefulness of immunosuppression for giant cell myocarditis. Am J Cardiol. 2008 Dec 1;102(11):1535-9. doi: 10.1016/j.amjcard.2008.07.041. Epub 2008 Sep 18. PMID 19026310